CLINICAL TRIAL: NCT04044872
Title: Single Institution Feasibility Study to Detect Radiation-Induced Cardiotoxicity in Receiving Thoracic Radiation Patients Using Hyperpolarized Carbon 13-Based Magnetic Resonance Spectroscopic Imaging
Brief Title: Hyperpolarized Carbon 13-Based Metabolic Imaging to Detect Radiation-Induced Cardiotoxicity
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: It has been terminated due to investigator decision to no longer pursue grant funding to support the study.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Prasanna Alluri, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU 2019-1099
Record Dates: First submitted 2019-07-10; First posted 2019-08-05 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Thoracic Cancer; Left Sided Breast Cancer
Keywords: Cardiotoxicity; Cardiac injury; Radiation induced heart disease (RIHD)
MeSH Terms: conditions — Unilateral Breast Neoplasms; Cardiotoxicity

STUDY DESIGN:
Intervention Model Description: [1-13C]pyruvate 0.1 mmol/kg dose will be injected twice at the time of imaging performed at baseline prior to standard of care radiation therapy and twice at 1 month or later after completion of standard of care radiation therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm:Diagnosing Cardiotoxicity when on Radiation therapy (Experimental)
  Interventions: Diagnostic Test: [1-13C]pyruvate along with MRI imaging

INTERVENTIONS:
Diagnostic Test: [1-13C]pyruvate along with MRI imaging — [1-13C]pyruvate: 0.1 mmol/kg dose will be injected at 5 mL/s followed by a 25 mL saline flush at 5 mL/s at the time of imaging performed at baseline (prior to radiation therapy), and 1 month after completion of radiation therapy.

SUMMARY:
Patients enrolled in the study will receive standard of care adjuvant or definitive breast, chest wall or thoracic radiation therapy.Cardiac mitochondrial dysfunction is a hallmark of radiation-induced cardiac injury. Reactive oxygen species (ROS) produced by ionizing radiation cause oxidation of mitochondrial proteins and alter oxidative phosphorylation and pyruvate metabolism(5). The goal of this study is to detect early changes in the mitochondrial metabolism in situ as a marker for subclinical radiation-induced cardiotoxicity.

DETAILED DESCRIPTION:
The global burden of cancer continues to rise with an incidence of 17.5 million cancer cases worldwide. Approximately 50% of all cancer patients receive radiation therapy as a component of their cancer care. While radiation therapy has demonstrable benefit in improving survival in patients with many types of malignancies, cardiotoxicity is a major concern in patients receiving chest radiotherapy. The rates of major coronary events increased by 7.4% per gray of mean heart dose; the increased risk was noted within the first 5 years of radiotherapy and persisted into the third decade after treatment. With improvements in multi-disciplinary care of cancer patients, the long-term survival in patients with thoracic malignancies continues to improve and radiation-induced heart disease (RIHD) is now a major source of morbidity and mortality in such patients.In this study, the investigators will enroll five female patients (18 years of age to 100 years of age) with left-sided breast cancer who underwent lumpectomy or mastectomy without tissue expander placement and will receive adjuvant standard-of-care breast or chest wall radiation therapy. They will undergo baseline magnetic resonance spectroscopic imaging with [1-13C]pyruvate injection and a proton MRI/spectroscopy scan prior to receipt of adjuvant radiation therapy. Post-treatment imaging will be performed within 3 months of completion of radiation treatments. This study will investigate whether non-invasive MRI scanning approaches will detect damage to the heart from left-sided radiation treatments before structural changes and mechanical functional deficits become apparent. A first-in-human clinical study to evaluate the effect of cardiotoxic chemotherapy on [1-13C]Pyruvate metabolism is currently ongoing at UT Southwestern (ClinicalTrials.gov Identifier: NCT03685175; PI: Dr. Vlad Zaha). The proposed study employs the same technology and approach to study radiation-induced cardiac toxicity. The study will also test the prognostic value of decreased myocardial mitochondrial pyruvate flux in predicting clinically significant radiation induced cardiotoxicity. Towards this goal, study will measure myocardial mechanical functional parameters, including left ventricular global longitudinal strain and left ventricular myocardial deformation using cardiac MRI and correlate these changes with [1-13C]lactate/ [13C]bicarbonate ratio. Previous studies have demonstrated that strain rate imaging by MRI is a sensitive technique for dose-dependent decrease in myocardial function after breast radiotherapy. Although this pilot study is restricted to breast cancer patients, successful demonstration of feasibility will allow extension of the study to all patients receiving thoracic radiation (such as patients receiving radiation therapy for lung cancer, esophageal cancer and thoracic lymphomas). The lack of reliable technologies for early detection of sub-clinical radiation-induced cardiotoxicity limits early intervention in such patients. Thus, identification of early cardiac changes induced by radiation therapy at a stage that offers potential for reversibility remains a major unmet need in cancer care.

Concerns for sexually active men and women: Women should not become pregnant and men should not father a baby while taking part in this study because we do not know how the study drugs/procedures could affect a man's sperm (for some drugs/procedures, the concern may be that the sperm might be affected and in some cases, drugs could being carried by the semen into the vagina and cause harm) or a fetus, if a woman becomes pregnant during the study. It is important that you talk to your study doctor about avoiding pregnancy during this study. If you think you might have become pregnant or if you believe your female partner has become pregnant while you are in this study, you must tell one of the study doctors right away so that management of the pregnancy and the possibility of stopping the study can be discussed.

ELIGIBILITY:
Inclusion Criteria:

1. Benign or malignant tumor of the breast (left-sided only) or thorax
2. Stage I to IV. If stage IV, patient must have life expectancy equal to or greater than 6 months
3. ECOG performance status 0-1
4. The patient must be deemed an appropriate candidate for standard of care radiation therapy
5. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   5.1 A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
   * Has not undergone a hysterectomy or bilateral oophorectomy; or
   * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

   5.2. A female of postmenopausal status is defined as patients over 60 or greater OR patients age 50-59 who meet the following criteria:
   * s/p bilateral oophorectomy, OR
   * with intact uterus without menses in the past 12 months OR,
   * with biochemical confirmation of post-menopausal status (estradiol in the menopausal range based on local laboratory criteria)
6. Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

1. Prior radiation involving the heart
2. Subjects may not be receiving any known cardiotoxic agents for the 6 months prior to the study and during the study
3. Diagnosis of connective tissue disorders, including systemic lupus erythematosis, scleroderma, or dermatomyositis
4. Patients with stage IV cancer with life expectancy of less than 6 months
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements
6. eGFR <30
7. Any contraindication to MRI (including, but not limited to metal implants and devices contraindicated at 3T, breast tissue expanders, non-MR compatible IV port, claustrophobia)
8. History of psychiatric or addictive disorders that would preclude obtaining informed consent
9. Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
To determine if radiation-induced cardiac injury causes myocardial mitochondrial dysfunction | at 1 month before the radiation
  To determine if radiation-induced cardiac injury causes myocardial mitochondrial dysfunction as measured by increase in [1-13C]lactate/ [13C]bicarbonate ratio and a decrease in [5-13C]glutamate formation in patients receiving radiotherapy to the thorax

SECONDARY OUTCOMES:
Determination of the prognostic value decreased of myocardial mitochondrial pyruvate flux in predicting clinically significant radiation induced cardiotoxicity. | At 1 month after the radiation
  As a secondary outcome, we will measure if decreased myocardial mitochondrial pyruvate flux results in changes in myocardial mechanical functional parameters. Towards this goal, we will measure myocardial mechanical functional parameters, including left ventricular global longitudinal strain and left ventricular myocardial deformation using cardiac MRI and correlate them with [1-13C] lactate/ [13C] bicarbonate ratio. Prior studies that cardiac MRI can detect changes in myocardial strain in patients who received whole breast radiotherapy for treatment of breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Prasanna Alluri, MD, PhD, Principal Investigator — UTSW Radiation Oncology
Locations (1):
- Department of Radiation Oncology; UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No